CLINICAL TRIAL: NCT02384538
Title: A Phase 2a, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study Comparing the Safety and Efficacy of ABT-981 to Placebo in Subjects With Erosive Hand Osteoarthritis
Brief Title: A Phase 2a Study Evaluating the Safety and Efficacy of ABT-981 in Patients With Erosive Hand Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M14-171; 2014-001096-31 (EudraCT Number)
Record Dates: First submitted 2015-03-05; First posted 2015-03-10 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-08-11 (Actual); Status verified 2017-07

CONDITIONS: Erosive Hand Osteoarthritis
Keywords: Osteoarthritis; Joint diseases; Musculoskeletal diseases; Rheumatic diseases; Arthritis; Osteoarthritis, Hand
MeSH Terms: conditions — Osteoarthritis; Joint Diseases; Musculoskeletal Diseases; Rheumatic Diseases; Arthritis | interventions — lutikizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo for ABT-981 every two weeks (Q2W) for 24 weeks.
  Interventions: Biological: Placebo for ABT-981
- ABT-981 (Experimental): ABT-981 200 mg every two weeks (Q2W) for 24 weeks.
  Interventions: Biological: ABT-981

INTERVENTIONS:
Biological: ABT-981 — ABT-981 administered by subcutaneous injection
  Other Names: lutikizumab
  Arms: ABT-981
Biological: Placebo for ABT-981 — Placebo for ABT-981 administered by subcutaneous injection
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled study to compare the safety and efficacy of ABT-981 to placebo in subjects with erosive hand osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 35 to 80.
2. Must fulfill 1990 American College of Rheumatology (ACR) hand osteoarthritis (OA) criteria
3. Must have radiographic evidence of erosive hand OA
4. Have one or more clinical signs and symptoms of active inflammation in at least three hand joints
5. Subject Assessment of Hand Pain Intensity in at least one hand is ≥ 6.

Exclusion Criteria:

1. Previous exposure to any anti-interleukin-1 treatment, to corticosteroids within 1 month prior to Screening, to intra-articular hyaluronic acid injection into hand joint(s) within 6 months prior to Screening, to any immunosuppressive biologic therapy within 1 month or 5 half-lives (whichever is longer) prior to the first dose of study drug, OR current use of immunosuppressive oral medications within 3 months or 5 half-lives (whichever is longer) prior to the first dose of study drug.
2. Absolute neutrophil count < 2,000 per mm3
3. Diagnosis of one or more of the following:

   * Fibromyalgia,
   * Inflammatory arthritis such as rheumatoid arthritis, peripheral seronegative spondyloarthropathy,
   * Psoriatic arthritis, psoriasis,
   * Microcrystalline (including gout and pseudo gout) arthritis affecting the hands,
   * Any OA of the hands due to an infectious origin or acute traumatic episode, secondary OA or OA linked to cartilage and bone dysplasia,
   * Other chronic painful syndromes that could interfere with assessment of pain at the hand(s).
4. Any uncontrolled medical illness or an unstable treatment or therapy.
5. Any reason that prohibits a subject to undergo an MRI.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc, Study Director — AbbVie

REFERENCES:
- [Derived] Kloppenburg M, Peterfy C, Haugen IK, Kroon F, Chen S, Wang L, Liu W, Levy G, Fleischmann RM, Berenbaum F, van der Heijde D, Bansal P, Wittoek R, Feng S, Fang Y, Saltarelli M, Medema JK, Levesque MC. Phase IIa, placebo-controlled, randomised study of lutikizumab, an anti-interleukin-1alpha and anti-interleukin-1beta dual variable domain immunoglobulin, in patients with erosive hand osteoarthritis. Ann Rheum Dis. 2019 Mar;78(3):413-420. doi: 10.1136/annrheumdis-2018-213336. Epub 2018 Dec 14. PMID 30552176

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 132 participants were randomized; 1 participant who was randomized to the ABT-981 treatment group did not receive a dose of study drug and was excluded from the analyses, for a total of 131 participants in the modified intent-to-treat population (mITT).
Period: Overall Study
Arm/Group | Placebo | ABT-981
Started | 67 | 64
Completed | 61 | 49
Not Completed | 6 | 15
Not completed — Adverse Event | 1 | 4
Not completed — Lack of Efficacy | 4 | 4
Not completed — Withdrew Consent | 0 | 4
Not completed — Other | 1 | 3

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population: all randomized participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | ABT-981 | Total
Number analyzed (Participants) | 67 | 64 | 131
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (7.325) | 65.7 (8.132) | 65.7 (7.700)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 53 | 111
  Male | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Australian/Canadian Hand Osteoarthritis Index (AUSCAN NR3.1) Pain Subdomain Score: Change From Baseline to Week 16
Description: The AUSCAN NR3.1 is a self-report measure composed of a battery of 15 questions assessing the three dimensions of pain (5 questions), joint stiffness (1 question) and physical function (9 questions) using an 11-box Numerical Rating Scale (NRS-11) from 0 (low) to 10 (high). The pain subdomain score ranges from 0 to 50; lower scores indicate better status. A decrease in the pain subdomain score represents improvement in status. Last Observation Carried Forward (LOCF): Missing responses were imputed by calculation based on the last nonmissing postbaseline component values.
Time Frame: Week 0 (Baseline), Week 16
Population: mITT population: all randomized participants who received at least 1 dose of study drug.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | ABT-981
Number analyzed (Participants) | 65 | 64
units on a scale | -10.74 [-15.433 to -6.045] | -9.22 [-13.798 to -4.645]
Statistical Analysis 1: Comparison: Placebo vs ABT-981; Test type: Other; p = 0.386, ANCOVA — P-value for test of difference in change from baseline between ABT-981 dose group and placebo is from an ANCOVA model with treatment group and country as the main factors and baseline as a covariate; LS Mean Difference = 1.52, 95% CI 2-sided [-1.944 to 4.990]

2. Secondary Outcome: Australian/Canadian Hand Osteoarthritis Index (AUSCAN NR3.1) Pain Subdomain Score: Change From Baseline to Each Visit
Description: The AUSCAN NR3.1 is a self-report measure composed of a battery of 15 questions assessing the three dimensions of pain (5 questions), joint stiffness (1 question) and physical function (9 questions) using an 11-box Numerical Rating Scale (NRS-11) from 0 (low) to 10 (high). The pain subdomain score ranges from 0 to 50; lower scores indicate better status. A decrease in the pain subdomain score represents improvement in status. LOCF: Missing responses were imputed by calculation based on the last nonmissing postbaseline component values.
Time Frame: Week 0 (Baseline) and Weeks 2, 4, 8, 12, 16, 20, and 26
Population: All participants in the mITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | ABT-981
Number analyzed (Participants) | 67 | 64
units on a scale
  Week 2: number analyzed (Participants) | 65 | 62
  Week 2 | -3.25 [-7.058 to 0.550] | -3.27 [-6.983 to 0.438]
  Week 4: number analyzed (Participants) | 65 | 64
  Week 4 | -5.01 [-9.144 to -0.885] | -4.26 [-8.280 to -0.237]
  Week 8: number analyzed (Participants) | 65 | 64
  Week 8 | -8.90 [-13.065 to -4.744] | -6.44 [-10.488 to -2.384]
  Week 12: number analyzed (Participants) | 65 | 64
  Week 12 | -8.31 [-12.593 to -4.030] | -5.64 [-9.809 to -1.469]
  Week 16: number analyzed (Participants) | 65 | 64
  Week 16 | -10.74 [-15.443 to -6.045] | -9.22 [-13.798 to -4.645]
  Week 20: number analyzed (Participants) | 65 | 64
  Week 20 | -7.28 [-11.969 to -2.591] | -8.37 [-12.941 to -3.807]
  Week 26: number analyzed (Participants) | 65 | 64
  Week 26 | -8.76 [-13.782 to -3.737] | -10.37 [-15.264 to -5.481]

3. Secondary Outcome: Australian/Canadian Hand Osteoarthritis Index (AUSCAN NR3.1) Physical Function Subdomain Score: Change From Baseline to Each Visit
Description: The AUSCAN NR3.1 is a self-report measure composed of a battery of 15 questions assessing the three dimensions of pain (5 questions), joint stiffness (1 question) and physical function (9 questions) using an 11-box Numerical Rating Scale (NRS-11) from 0 (low) to 10 (high). The physical function subdomain score ranges from 0 to 90; lower scores indicate better status. A decrease in the physical function subdomain score represents improvement in status. LOCF: Missing responses were imputed by calculation based on the last nonmissing postbaseline component values.
Time Frame: Week 0 (Baseline) and Weeks 2, 4, 8, 12, 16, 20, and 26
Population: All participants in the mITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | ABT-981
Number analyzed (Participants) | 67 | 64
units on a scale
  Week 2: number analyzed (Participants) | 65 | 62
  Week 2 | -6.23 [-13.098 to 0.630] | -4.79 [-11.440 to 1.861]
  Week 4: number analyzed (Participants) | 65 | 64
  Week 4 | -8.43 [-15.879 to -0.974] | -7.04 [-14.249 to 0.177]
  Week 8: number analyzed (Participants) | 65 | 64
  Week 8 | -14.25 [-21.729 to -6.763] | -8.97 [-16.211 to -1.725]
  Week 12: number analyzed (Participants) | 65 | 64
  Week 12 | -12.54 [-20.140 to -4.947] | -8.53 [-15.887 to -1.182]
  Week 16: number analyzed (Participants) | 65 | 64
  Week 16 | -17.18 [-24.938 to -9.431] | -14.64 [-22.142 to -7.133]
  Week 20: number analyzed (Participants) | 65 | 64
  Week 20 | -11.50 [-19.415 to -3.584] | -12.53 [-20.189 to -4.867]
  Week 26: number analyzed (Participants) | 65 | 64
  Week 26 | -14.25 [-22.523 to -5.978] | -16.39 [-24.402 to -8.388]
Statistical Analysis 1: Comparison: Placebo vs ABT-981; Week 16; Test type: Other; p = 0.383, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 2.55, 95% CI 2-sided [-3.214 to 8.308]

4. Secondary Outcome: Australian/Canadian Hand Osteoarthritis Index (AUSCAN NR3.1) Stiffness Subdomain Score: Change From Baseline to Each Visit
Description: The AUSCAN NR3.1 is a self-report measure composed of a battery of 15 questions assessing the three dimensions of pain (5 questions), joint stiffness (1 question) and physical function (9 questions) using an 11-box Numerical Rating Scale (NRS-11) from 0 (low) to 10 (high). The stiffness subdomain score ranges from 0 to 10; lower scores indicate better status. A decrease in the stiffness subdomain score represents improvement in status. LOCF: Missing responses were imputed by calculation based on the last nonmissing postbaseline component values.
Time Frame: Week 0 (Baseline) and Weeks 2, 4, 8, 12, 16, 20, and 26
Population: All participants in the mITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | ABT-981
Number analyzed (Participants) | 67 | 64
units on a scale
  Week 2: number analyzed (Participants) | 65 | 62
  Week 2 | -0.74 [-1.692 to 0.215] | -0.96 [-1.877 to -0.036]
  Week 4: number analyzed (Participants) | 65 | 64
  Week 4 | -0.98 [-1.937 to -0.028] | -1.24 [-2.163 to -0.321]
  Week 8: number analyzed (Participants) | 65 | 64
  Week 8 | -1.51 [-2.535 to -0.493] | -1.43 [-2.412 to -0.441]
  Week 12: number analyzed (Participants) | 65 | 64
  Week 12 | -1.65 [-2.706 to -0.599] | -1.23 [-2.244 to -0.211]
  Week 16: number analyzed (Participants) | 65 | 64
  Week 16 | -1.76 [-2.885 to -0.633] | -1.61 [-2.695 to -0.522]
  Week 20: number analyzed (Participants) | 65 | 64
  Week 20 | -1.34 [-2.515 to -0.169] | -1.85 [-2.986 to -0.722]
  Week 26: number analyzed (Participants) | 65 | 64
  Week 26 | -1.94 [-3.017 to -0.859] | -2.45 [-3.492 to -1.410]
Statistical Analysis 1: Comparison: Placebo vs ABT-981; Week 16; Test type: Other; p = 0.719, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 0.15, 95% CI 2-sided [-0.677 to 0.979]

5. Secondary Outcome: Australian/Canadian Hand Osteoarthritis Index (AUSCAN NR3.1) Total Score: Change From Baseline to Each Visit
Description: The AUSCAN NR3.1 is a self-report measure composed of a battery of 15 questions assessing the three dimensions of pain (5 questions), joint stiffness (1 question) and physical function (9 questions) using an 11-box Numerical Rating Scale (NRS-11) from 0 (low) to 10 (high). The total score ranges from 0 to 150; lower scores indicate better status. A decrease in the total score represents improvement in status. LOCF: Missing responses were imputed by calculation based on the last nonmissing postbaseline component values.
Time Frame: Week 0 (Baseline) and Weeks 2, 4, 8, 12, 16, 20, and 26
Population: All participants in the mITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | ABT-981
Number analyzed (Participants) | 67 | 64
units on a scale
  Week 2: number analyzed (Participants) | 65 | 62
  Week 2 | -10.01 [-21.037 to 1.019] | -8.85 [-19.545 to 1.835]
  Week 4: number analyzed (Participants) | 65 | 64
  Week 4 | -14.06 [-26.185 to -1.930] | -12.18 [-23.928 to -0.439]
  Week 8: number analyzed (Participants) | 65 | 64
  Week 8 | -24.52 [-36.660 to -12.373] | -16.65 [-28.406 to -4.886]
  Week 12: number analyzed (Participants) | 65 | 64
  Week 12 | -22.29 [-34.714 to -9.873] | -15.15 [-27.181 to -3.124]
  Week 16: number analyzed (Participants) | 65 | 64
  Week 16 | -29.37 [-42.469 to -16.264] | -25.12 [-37.808 to -12.429]
  Week 20: number analyzed (Participants) | 65 | 64
  Week 20 | -19.68 [-32.894 to -6.458] | -22.33 [-35.128 to -9.526]
  Week 26: number analyzed (Participants) | 65 | 64
  Week 26 | -24.73 [-38.636 to -10.820] | -28.99 [-42.461 to -15.523]
Statistical Analysis 1: Comparison: Placebo vs ABT-981; Week 16; Test type: Other; p = 0.387, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 4.25, 95% CI 2-sided [-5.448 to 13.945]

6. Secondary Outcome: Participant Assessment of Index Hand Pain Intensity Using Numeric Rating Scale (NRS-11): Change From Baseline to Each Visit
Description: Participants rated the pain intensity of each hand during the previous 48 hours using an 11-point scale (NRS-11). The change from baseline to each visit in NRS-11 in the index hand (the hand with the most disease) are presented. Scores range from 0 to 10 points, with higher scores indicating greater pain intensity. A decrease in the NRS-11 score represents a decrease in pain intensity.
Time Frame: Week 0 (Baseline) and Weeks 2, 4, 8, 12, 16, 20, and 26
Population: All participants in the mITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | ABT-981
Number analyzed (Participants) | 67 | 64
units on a scale
  Week 2: number analyzed (Participants) | 65 | 62
  Week 2 | -0.62 [-1.550 to 0.320] | -0.69 [-1.613 to 0.228]
  Week 4: number analyzed (Participants) | 65 | 63
  Week 4 | -1.18 [-2.163 to -0.195] | -1.06 [-2.025 to -0.088]
  Week 8: number analyzed (Participants) | 63 | 58
  Week 8 | -2.40 [-3.339 to -1.465] | -1.74 [-2.660 to -0.814]
  Week 12: number analyzed (Participants) | 61 | 53
  Week 12 | -1.65 [-2.434 to -0.875] | -0.81 [-1.629 to 0.010]
  Week 16: number analyzed (Participants) | 61 | 51
  Week 16 | -2.05 [-3.085 to -1.017] | -1.60 [-2.626 to -0.578]
  Week 20: number analyzed (Participants) | 57 | 49
  Week 20 | -1.61 [-2.749 to -0.477] | -1.75 [-2.892 to -0.612]
  Week 26: number analyzed (Participants) | 60 | 50
  Week 26 | -2.02 [-3.132 to -0.901] | -2.52 [-3.620 to -1.415]
Statistical Analysis 1: Comparison: Placebo vs ABT-981; Week 16; Test type: Other; p = 0.281, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 0.45, 95% CI 2-sided [-0.373 to 1.272]

7. Secondary Outcome: Patient Global Assessment of Hand Osteoarthritis (OA) Status by NRS-11: Change From Baseline to Each Visit
Description: Participants were asked how much they were affected by hand OA by responding to the question "Considering all the ways your hand OA affects you, how have you been during the last 48 hours?" using an 11-point scale (NRS-11). Scores range from 0 to 10 points, with higher scores indicating greater effect of hand OA on the participant. A decrease in the NRS-11 score represents an improvement the effect of hand OA on the participant.
Time Frame: Week 0 (Baseline) and Weeks 2, 4, 8, 12, 16, 20, and 26
Population: All participants in the mITT population.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Placebo | ABT-981
Number analyzed (Participants) | 67 | 64
units on a scale
  Week 2: number analyzed (Participants) | 65 | 62
  Week 2 | -0.52 [-1.399 to 0.351] | -0.54 [-1.403 to 0.316]
  Week 4: number analyzed (Participants) | 65 | 63
  Week 4 | -1.31 [-2.277 to -0.335] | -1.13 [-2.083 to -0.176]
  Week 8: number analyzed (Participants) | 63 | 58
  Week 8 | -1.85 [-2.740 to -0.952] | -1.20 [-2.080 to -0.324]
  Week 12: number analyzed (Participants) | 61 | 53
  Week 12 | -1.78 [-2.567 to -0.993] | -1.17 [-1.997 to -0.348]
  Week 16: number analyzed (Participants) | 61 | 51
  Week 16 | -2.20 [-3.225 to -1.185] | -1.69 [-2.697 to -0.677]
  Week 20: number analyzed (Participants) | 57 | 49
  Week 20 | -1.73 [-2.836 to -0.627] | -1.77 [-2.879 to -0.666]
  Week 26: number analyzed (Participants) | 60 | 50
  Week 26 | -2.00 [-3.133 to -0.874] | -2.35 [-3.465 to -1.236]
Statistical Analysis 1: Comparison: Placebo vs ABT-981; Week 16; Test type: Other; p = 0.212, ANCOVA — [p-value comment as in outcome 1, analysis 1]; LS Mean Difference = 0.52, 95% CI 2-sided [-0.300 to 1.336]

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 70 days after the last dose of study drug (up to 34 weeks).
Description: TEAEs and TESAEs are defined as any AE or SAE that begins on or after the first dose of study drug, up to 70 days after the last dose of study drug.
Arm/Group | Placebo | ABT-981
Serious Adverse Events (participants affected / at risk) | 2/67 | 2/64
Other Adverse Events (participants affected / at risk) | 45/67 | 49/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=67) | ABT-981 (N=64)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 | 0
FAECES DISCOLOURED (Gastrointestinal disorders) | 0 | 1
HAEMOGLOBIN DECREASED (Investigations) | 0 | 1
INVASIVE BREAST CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=67) | ABT-981 (N=64)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 | 6
DIARRHOEA (Gastrointestinal disorders) | 6 | 4
NAUSEA (Gastrointestinal disorders) | 2 | 8
FATIGUE (General disorders) | 0 | 4
INJECTION SITE ERYTHEMA (General disorders) | 0 | 7
INJECTION SITE RASH (General disorders) | 3 | 7
INJECTION SITE REACTION (General disorders) | 3 | 7
PAIN (General disorders) | 4 | 0
NASOPHARYNGITIS (Infections and infestations) | 17 | 13
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 4
FALL (Injury, poisoning and procedural complications) | 3 | 4
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6 | 4
BACK PAIN (Musculoskeletal and connective tissue disorders) | 11 | 3
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 4 | 3
DIZZINESS (Nervous system disorders) | 4 | 4
HEADACHE (Nervous system disorders) | 17 | 10
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 5 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.